CLINICAL TRIAL: NCT00343473
Title: Novel Diagnostics With Optical Coherence Tomography: Imaging of the Anterior Eye
Brief Title: Novel Diagnostics With Optical Coherence Tomography: Imaging the Anterior Eye
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: s17-00039; R01EY011289-15 (NIH); NCT00343746 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-23 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Fuch's Dystrophy; Corneal Disorders; Prior Surgery
Keywords: Fuch's dystrophy; corneal disorders; cornea; lasik; refractive surgery
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to evaluate the optical coherence tomography (OCT), to image diseases of the eye. OCT may be useful for the early diagnosis and monitoring of a variety of diseases involving the eye, such as Fuch's Dystrophy (type of eye disease) and retinal damage (eye diseases in the back of the eye) due to diabetes.

DETAILED DESCRIPTION:
The purpose of this research is to evaluate the optical coherence tomography (OCT), to image diseases of the eye. OCT may be useful for the early diagnosis and monitoring of a variety of diseases involving the eye, such as Fuch's Dystrophy (type of eye disease) and retinal damage (eye diseases in the back of the eye) due to diabetes. OCT may also be useful for assessing contact lens and surgical procedures, such as LASIK (type of ophthalmic surgical procedure). The OCT is Food and Drug Administration (FDA) approved. The ultra high OCT is a non-significant risk device (it does not present a possible serious risk to your health, your safety, or your welfare) that has not been approved by the FDA. This study will also be conducted at the Massachusetts Institute of Technology and Tufts-New England Medical Center New England Eye Center in Massachusetts

ELIGIBILITY:
Inclusion Criteria: Female Subjects who are pregnant or breastfeeding will be included (no risks to fetus).

Normals: Normal appearing cornea, no history of corneal trauma, surgery or disease, no historical or current contact lens wear. Thirty subjects from 6 different age groups (> 18 yrs; 20-30 yrs; 30-40 yrs; 40-50 yrs; 50-60 yrs; > 60 yrs) will be recruited to determine the normal variations in anterior eye structure.

LASIK patients: to participate as a LASIK patient, the subject is previously normal but may have worn contact lenses, and is scheduled to undergo LASIK.

Contact lens wearers: to participate as a contact lens wearer the patient otherwise fulfills all criteria specified for normalcy, with the exception of contact lens wear.

Fuchs' dystrophy patients: Fuchs' Dystrophy is characterized by guttata and clinically significant corneal edema, with a corneal thickness of >700 microns, and/or reduced visual acuity in the morning which improves over the course of the day.

Diabetic patients: for diabetic patients are specified in the posterior segment imaging section.

-

Exclusion Criteria:Subjects will be excluded from the study if their media are opaque, or if they are unwilling or unable to participate in the study.

If participants choose they may also participate in other imaging research protocols. No risk is associated if entering multiple imaging protocols, while being a participant in this research study.

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will range form 18 years to 90 years. Gender can be male or female. Will include 100 normals and 100 diseased patients that include diabetic retinopathy, macular degeneration, and glaucoma.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Novel Diagnostics With Optical Coherence Tomography: Imaging the Anterior Eye | 2 years
  The purpose of this research is to evaluate the optical coherence tomography (OCT), to image diseases of the eye. OCT may be useful for the early diagnosis and monitoring of a variety of diseases involving the eye, such as Fuch's Dystrophy (type of eye disease) and retinal damage (eye diseases in the back of the eye) due to diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Chaim Wollstein, MD, Principal Investigator — NYU Langone Health; Ian Conner, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - New York University School of Medicine, New York, New York
  - University of Pittsburgh UPMC Eye Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Christopoulos V, Kagemann L, Wollstein G, Ishikawa H, Gabriele ML, Wojtkowski M, Srinivasan V, Fujimoto JG, Duker JS, Dhaliwal DK, Schuman JS. In vivo corneal high-speed, ultra high-resolution optical coherence tomography. Arch Ophthalmol. 2007 Aug;125(8):1027-35. doi: 10.1001/archopht.125.8.1027. PMID 17698748